CLINICAL TRIAL: NCT06345209
Title: A Prospective, Multicenter, Randomized Controlled, Noninferiority Clinical Trial Evaluating the Safety and Efficacy of Sirolimus-coated Coronary Balloon Dilatation Catheter for the Treatment of De Novo Coronary Artery Small Vessel Lesions.
Brief Title: Efficacy and Safety of Sirolimus-coated Coronary Balloon Dilatation Catheter for Coronary Small Vessels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM-D19
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Sirolimus-coated Coronary Balloon Dilatation Catheter
  Interventions: Device: Sirolimus-coated Coronary Balloon Dilatation Catheter
- Control Group (Active Comparator): Drug Eluting Balloon Catheter
  Interventions: Device: Drug-coated Coronary Balloon Dilatation Catheter

INTERVENTIONS:
Device: Sirolimus-coated Coronary Balloon Dilatation Catheter — During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using the Sirolimus-coated Coronary Balloon Dilatation Catheter in the test group, subsequently completing the remaining procedure
  Arms: Test Group
Device: Drug-coated Coronary Balloon Dilatation Catheter — During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using the Drug-coated Coronary Balloon Dilatation Catheter in the test group, subsequently completing the remaining procedure
  Arms: Control Group

SUMMARY:
To evaluate the safety and efficacy of a sirolimus-coated coronary balloon dilatation catheter for the treatment of small vessel lesions of primary coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited
2. Diagnosed with stable or unstable angina, old myocardial infarction, or asymptomatic myocardial ischemia
3. Suitable for balloon angioplasty
4. Be able to understand the purpose of the trial, be willing to cooperate in the follow-up, and voluntarily sign an informed consent form.
5. Primary coronary small vessel lesions with a visual lesion length of ≤36mm and a visual lesion diameter of ≥2.00mm and ≤2.75mm
6. Target lesions with ≥70% or ≥50% diameter stenosis with evidence of ischemia before interventional therapy
7. Residual stenosis of ≤30% visualized after pre-interventional dilatation of the target lesion without type C or higher entrapment
8. In the presence of multiple lesions requiring treatment, one of the lesions that meets the requirements should be selected as the target lesion, and the non-target lesion should be in a different vascular branch from the target lesion.
9. Patients with at most two non-target lesions requiring simultaneous treatment, and the non-target lesion should undergo interventional therapy before the target lesion, and there are no serious complications after treatment.

Exclusion Criteria:

Patients who had a myocardial infarction within 7 days before enrollment (2) Patients with cardiogenic shock (3) Patients with renal insufficiency (eGFR < 30 ml/min) or vital organ failure (4) Patients with known allergy or intolerance to contrast media or to rapamycin, paclitaxel and/or their analogs (5) Patients with hematologic disorders, or contraindications to anticoagulant/antiplatelet agents, or intolerance to aspirin or clopidogrel (6) Patients with severe valvular heart disease or who have undergone heart transplantation (7) Patients who are not suitable for coronary artery bypass graft surgery (CABG) (8) Patients with congestive heart failure or NYHA class IV (9) Patients who have had a stroke within 6 months prior to enrollment, or have a history of gastrointestinal bleeding or active gastric ulcers, or who have been determined by the investigator to have a bleeding constitution (10) Patients with a life expectancy of less than 1 year (11) Pregnant or lactating females (12) Patients who are participating in clinical trials of other drugs or medical devices (13) Patients who, in the opinion of the investigator, are not suitable for enrollment for other reasons.

(14) Totally occluded (TIMI grade 0) lesions (15) Presence of coronary artery spasm without significant stenosis (16) Unprotected left main stem lesions (17) Patients with a bifurcation lesion (branch diameter ≥2.00 mm) as the target lesion (18) Patients with target lesions that are severely tortuous (preventing smooth catheter passage) or severely calcified (19) Patients with secondary stenosis caused by pre-dilatation of the target lesion (20) Patients with a well-defined thrombus in the target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Late luminal loss (LLL) | 9 months after procedure
  Late luminal loss (LLL) within the target lesion segment at 9 months postoperatively

SECONDARY OUTCOMES:
Device success rate | Immediately after PTCA
  Successful delivery and dilatation of the drug-coating balloon catheter across lesion, and target lesion residual stenosis≤30% (visual inspection) without additional interventional treatment.